CLINICAL TRIAL: NCT01733186
Title: Evaluation of Safety and Exploratory Efficacy of CARTISTEM®, a Cell Therapy Product for Articular Cartilage Defects: A Phase I/IIa Clinical Trial in Patients With Focal, Full-thickness Grade 3-4 Articular Cartilage Defects of the Knee
Brief Title: Evaluation of Safety and Exploratory Efficacy of CARTISTEM®, a Cell Therapy Product for Articular Cartilage Defects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medipost, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-0201-01
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Degeneration Articular Cartilage Knee
Keywords: human umbilical cord blood-derived mesenchymal stem cells; MSC; cartilage lesion; cartilage defect; degenerative arthritis; stem cell implantation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CARTISTEM® (Experimental): Drug name and ingredients: CARTISTEM [allogeneic-unrelated, umbilical cord blood-derived mesenchymal stem cells, ex vivo cultured, combined with sodium hyaluronate] Dosage: Administer 0.5 mL of the combination product per cm^2 of the cartilage defect
  Interventions: Biological: CARTISTEM®

INTERVENTIONS:
Biological: CARTISTEM®
  Other Names: human umbilical cord blood-derived mesenchymal stem cells

SUMMARY:
The purpose of this study is to determine whether CARTISTEM, a cell therapeutic product, is safe and effective in the treatment of articular cartilage defects of the knee as a result of ageing, trauma, or degenerative diseases.

DETAILED DESCRIPTION:
Conventional treatment modalities have not been able to provide complete and sustained resolution of symptoms following damage to the articular cartilage. Despite the numerous techniques available today, complete healing of damaged or defective cartilage or consistent reproduction of normal hyaline cartilage does not occur, and continuous drug administration or secondary surgeries are common.

Research in mesenchymal stem cells has had a rapid acceleration over the past decade and MSC-based therapy has become one of the objects of investigation for a new branch of medicine termed regenerative medicine. This emerging technology shows great promise for producing transplantable cartilage constructs to restore the function of degenerated joints.

CARTISTEM®, a combination of human umbilical cord blood-derived mesenchymal stem cells and sodium hyaluronate, is intended to be used as a single-dose cellular therapeutic agent for cartilage regeneration in human subjects with cartilage defects of the knee as a result of ageing, trauma, or degenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an intended- to- treat single focal, full-thickness cartilage defect (ICRS [International Cartilage Repair Society] Grade 3 or 4) of the knee as a result of ageing, trauma, or degenerative diseases.
* Age ≥ 18 years old
* Size of the articular cartilage lesion is ≥ 2 cm2
* Swelling, tenderness and active range of motion ≤ Grade II
* Joint pain : 20-mm - 60-mm on VAS (Visual Analog Scale) at the time of Screening
* Appropriate blood coagulation, kidney and liver function laboratory parameters: PT(INR) < 1.5, APTT <1.5×control Creatinine ≤ 2.0 mg/dL Albumin ≤ trace in urine dipstick test Bilirubin ≤ 2.0 mg/dL, AST/ALT ≤ 100 IU/L
* Ligament instability ≤ Grade II
* Lower extremity alignment within 5 degrees of the neutral weight bearing axis
* No meniscal surgery within the past 3 months and more than 5mm of meniscal rim remaining
* Ability and willingness to fully participate in the post-operative rehabilitation program
* Subject is informed of the investigational nature of this study, voluntarily agrees to participate in the study, and signs an IRBapproved informed consent prior to performing any of the screening procedures
* Body Mass Index (BMI) ≤ 35 kg/m2

Exclusion Criteria:

* Patients who have been treated previously and are asymptomatic
* Avascular necrosis/ osteonecrosis
* Autoimmune or inflammatory joint disease
* History of infection within the past 6 weeks
* Surgery or radiation therapy within the past 6 weeks
* Serious medical co-morbidities, which would otherwise contraindicate surgery, as determined by the investigator
* Currently pregnant or nursing
* Psychotic diseases, epilepsy, or any history of such diseases
* Current abuse of alcohol (> 10 drinks weekly) and/or regular exposure to other substances of abuse, currently an active smoker
* Chronic inflammatory articular diseases such as rheumatoid arthritis
* Enrolled in any other clinical trials within the past 4 weeks
* Administered immunosuppressants such as Cyclosporin A or azathioprine within the past 6 weeks
* Ligament instability > Grade II
* Uncorrected significant lower extremity malalignment (i.e. > 5 degrees)
* (sub-) Total meniscectomy (<5mm rim remaining)
* Corticosteroid or viscosupplementation injection to the affected knee in the past 3 months
* Principal investigator considers inappropriate for the clinical trial due to any reasons other than those listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Cole, MD, Principal Investigator — Cartilage Restoration Center, Rush University Medical Center; Andreas H Gomoll, MD, Principal Investigator — Cartilage Repair Center, Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Cartilage Restoration Center; RUSH University Medical Center, Chicago, Illinois
  - Cartilage Repair Center; Brigham and Women's Hospital, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study to Compare the Efficacy and Safety of Cartistem® and Microfracture in Patients With Knee Articular Cartilage Injury or Defect — http://clinicaltrials.gov/ct2/show/NCT01041001?term=cartistem&rank=2

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose A Cohort: Drug name and ingredients: CARTISTEM [allogeneic-unrelated, umbilical cord blood-derived mesenchymal stem cells, ex vivo cultured, combined with sodium hyaluronate] Dosage: Administer 0.5 mL of the combination product per cm^2 of the cartilage defect
  Cartilage defect size range: 2 to 5 cm2 (Dose A)
  CARTISTEM®
- Dose B Cohort: Drug name and ingredients: CARTISTEM [allogeneic-unrelated, umbilical cord blood-derived mesenchymal stem cells, ex vivo cultured, combined with sodium hyaluronate] Dosage: Administer 0.5 mL of the combination product per cm^2 of the cartilage defect
  Cartilage defect size range: above 5 cm2 (Dose B)
  CARTISTEM®
Period: Overall Study
Arm/Group | Dose A Cohort | Dose B Cohort
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose A Cohort | Dose B Cohort | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (8.2) | 39.7 (8.0) | 38.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (4.1) | 26.6 (4.5) | 27.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: IKDC Score
Description: Subjects underwent a self-assessment of knee function using the IKDC (International Knee Documentation Committee Assessment)subjective knee evaluation before and after the administration of the IP. The assessment is designed to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment. The possible score ranges from 0 to 100, where 100 = no limitation with daily or sporting activities and the absence of symptoms.
  The IKDC assessment was performed before IP administration and at Months 12 after IP administration in an exploratory fashion. The IKDC score from the Month 12 visit was used as a primary indicator of the post operative change.
  The outcome was presented with the post-operative change amount from the baseline.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose A Cohort | Dose B Cohort
Number analyzed (Participants) | 6 | 6
score on a scale | 32.0 (27.7) | 25.5 (18.9)

2. Secondary Outcome: VAS
Description: Subjects underwent a self-assessment of joint pain using the 100-mm VAS (Visual Analogue Scale) before and at Months 12 and 24 after IP (investigational product) administration. Higher values represent worse joint pain. Use of NSAIDs and any other analgesics had to be discontinued for 48 hours and 24 hours, respectively, prior to the 100 mm VAS evaluation. The outcome was presented with the post-operative change amount at Months 12 and 24 from the baseline.
  100-mm VAS scores range from 0 to 100. Higher values represent worse joint pain.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose A Cohort | Dose B Cohort
Number analyzed (Participants) | 6 | 6
score on a scale
  12 MONTHS | -23.8 (22.9) | -12.5 (31.5)
  24 MONTHS | -31.7 (18.0) | -11.3 (30.2)

3. Secondary Outcome: Lysholm Score
Description: The Lysholm knee scoring scale is a self-assessment that rates the severity of common complaints related to knee problems, such as pain, swelling, abnormal sensations, and ability to squat or climb stairs. The possible score ranges from 0 to 100, where 100 = no symptoms or disability. Scores are categorized as excellent (95 to 100), good (84 to 94), fair (65 to 83), and poor (≤64). Subjects underwent a self-assessment of knee function using the Lysholm score before IP administration and at Months 12 and 24 after IP administration. The outcome was presented with the post-operative change amount at Months 12 and 24 from the baseline.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose A Cohort | Dose B Cohort
Number analyzed (Participants) | 6 | 6
score on a scale
  12 MONTHS | 26.7 (20.5) | 22.5 (18.3)
  24 MONTHS | 32.0 (20.9) | 10.2 (13.0)

4. Secondary Outcome: KOOS Score
Description: The Knee Injury and Osteoarthritis Outcome score (KOOS) knee survey is a self assessment of knee function and knee-related quality of life (QOL). Subjects responded to each question regarding knee-related symptoms, swelling, pain, impaired function, or changes in QOL with 1 of 5 possible answers that range from "never/not at all" to "always/extremely." The possible score for each parameter ranges from 0 to 100, where 0=extreme problems and 100=no problems. Subjects completed the KOOS knee survey before IP (investigational product) administration and at Month 24 after IP administration. The outcome was presented with the post-operative change amount at Month 24 from the baseline.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose A Cohort | Dose B Cohort
Number analyzed (Participants) | 6 | 6
score on a scale
  ADL (24 MONTHS) | 28.2 (25.7) | 12.3 (19.2)
  PAIN (24 MONTHS) | 23.6 (24.3) | 15.8 (13.1)
  QOL (24 MONTHS) | 50.0 (36.4) | 19.8 (24.2)
  SPORTS (24 MONTHS) | 39.2 (37.2) | 36.7 (31.9)
  SYMPTOM (24 MONTHS) | 24.4 (19.9) | 8.3 (12.3)

5. Secondary Outcome: IKDC Score
Description: Subjects underwent a self-assessment of knee function using the IKDC subjective knee evaluation before and after the administration of the IP. The assessment is designed to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment. The possible score ranges from 0 to 100, where 100 = no limitation with daily or sporting activities and the absence of symptoms. The IKDC assessment was performed before IP administration and at Month 24 after IP administration in an exploratory fashion. The outcome was presented with the post-operative change amount at Month 24 from the baseline.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose A Cohort | Dose B Cohort
Number analyzed (Participants) | 6 | 6
score on a scale | 41.2 (25.8) | 27.5 (20.9)

ADVERSE EVENTS:
Time Frame: 24 months
Description: General safety was evaluated via the following assessments: adverse events (AEs), routine clinical laboratory tests (hematology, clinical chemistry, and urinalysis), thrombin generation (prothrombin time and activated partial thromboplastin time [aPTT]), immunogenicity tests (T cell subset), vital signs, physical examinations, and magnetic resonance imaging (MRI) for tumorigenicity.
Arm/Group | Dose A Cohort | Dose B Cohort
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose A Cohort (N=6) | Dose B Cohort (N=6)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (6)
bone marrow oedema (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
blood pressure increased (Investigations) | 1 (1) | 0 (0)
nuclear magnetic resonance imaging abnormal (Investigations) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (9)
joint effusion (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
muscle atrophy (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
joint crepitation (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
joint lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
plica syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
prehypertension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT01733186/Prot_SAP_000.pdf